CLINICAL TRIAL: NCT00157755
Title: Gastric Stimulation for Vomiting, Nausea and Related Symptoms Associated With Gastroparesis Using Enterra® Gastric Stimulation System
Brief Title: Enterra Therapy Clinical Study (Gastric Stimulation for Gastroparesis)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Darin Lerew, Sr. Clinical Manager, Medtronic Neuromodulation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NDHF0025-70006
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2009-12

CONDITIONS: Gastroparesis
Keywords: Nausea and Vomiting
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Device: Enterra Therapy — Gastric electrical stimulation using Enterra Therapy.

SUMMARY:
This study is to evaluate the safety and effectiveness of gastric stimulation in the reduction of nausea and vomiting in patients with gastroparesis using an approved Humanitarian device. There are two cohorts in this study based on etiology, one for diabetic and one for idiopathic.

A maximum of 150 patients (75 diabetic and 75 idiopathic) from up to 15 centers in the United States will be followed closely for twelve months and then once a year after that until the study closes.

If you are someone suffering with symptoms of gastroparesis despite trying oral medications, you may be eligible to participate in a clinical study using a surgically implanted gastric stimulator.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age
* Diagnosed with gastroparesis due to diabetes or an unknown cause (idiopathic)
* Have tried prokinetic (help the stomach empty quicker) and antiemetic (help decrease symptoms of nausea and vomiting) medications for a minimum of one month, unless you're unable to take these types of medications
* Have symptoms of gastroparesis that have required treatment for at least one year
* Experience at least 7 episodes of vomiting during a seven consecutive day period on a 28-day diary
* Willing and able to completely and accurately fill out a diary and questionnaires throughout the study
* Have gastric retention of greater than 10% at four hours, or greater than 60% at two hours (if unable to complete the four-hour test) on a Gastric Emptying Test (GET)

Exclusion Criteria:

* Gastroparesis caused by a specific diagnosed illness other than diabetes
* Current eating disorder or diagnosed swallowing disorder
* Previous stomach surgeries
* Taking narcotic pain-relievers daily for abdominal pain
* Diagnosed with drug or alcohol dependency within 1 year before the study
* Life expectancy less than one year
* Have other implantable devices such as pacemakers
* Pregnancy or planned pregnancy
* Plan to receive diathermy treatment
* Have had radiation therapy of the upper abdomen
* Plan on having an MRI performed
* Currently participating in another investigational device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2002-06; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darin R Lerew, PhD, Study Director — Medtronic
Locations (6):
- United States (6):
  - Contact Medtronic for exact location, San Francisco, California
  - Contact Medtronic for exact location, Washington D.C., District of Columbia
  - Contact Medtronic for exact location, Anderson, Indiana
  - Contact Medtronic for exact location, Kansas City, Kansas
  - Contact Medtronic for exact location, Louisville, Kentucky
  - Contact Medtronic for exact location, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] McCallum RW, Snape W, Brody F, Wo J, Parkman HP, Nowak T. Gastric electrical stimulation with Enterra therapy improves symptoms from diabetic gastroparesis in a prospective study. Clin Gastroenterol Hepatol. 2010 Nov;8(11):947-54; quiz e116. doi: 10.1016/j.cgh.2010.05.020. Epub 2010 Jun 9. PMID 20538073

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic: ON First, Then OFF: This group contains subjects that were enrolled and analyzed as part of the diabetic cohort. During the crossover phase of the study, this subject had the device ON for three months, followed by device OFF for three months.
- Diabetic: OFF First, Then ON: This group contains subjects that were enrolled and analyzed as part of the diabetic cohort. During the crossover phase of the study, this subject had the device OFF for three months, followed by device ON for three months.
- Diabetic: Not Randomized: This group contains subjects that were enrolled and analyzed as part of the diabetic cohort. These subjects exited the study prior to randomization at 1.5 months.
- Idiopathic: ON First, Then OFF: This group contains subjects that were enrolled and analyzed as part of the idiopathic cohort. During the crossover phase of the study, this subject had the device ON for three months, followed by device OFF for three months.
- Idiopathic: OFF First, Then ON: This group contains subjects that were enrolled and analyzed as part of the idiopathic cohort. During the crossover phase of the study, this subject had the device OFF for three months, followed by device ON for three months.
- Idiopathic: Not Randomized: This group contains subjects that were enrolled and analyzed as part of the idiopathic cohort. These subjects exited the study prior to randomization at 1.5 months.
Period: Overall Study
Arm/Group | Diabetic: ON First, Then OFF | Diabetic: OFF First, Then ON | Diabetic: Not Randomized | Idiopathic: ON First, Then OFF | Idiopathic: OFF First, Then ON | Idiopathic: Not Randomized
Started | 26 | 19 | 10 | 15 | 12 | 5
Completed | 24 (Subjects finished 12-month follow-up.) | 15 (Subjects finished 12-month follow-up.) | 3 (Subjects finished 12-month follow-up.) | 11 (Subjects finished 12-month follow-up.) | 10 (Subjects finished 12-month follow-up.) | 0 (Subjects finished 12-month follow-up.)
Not Completed | 2 | 4 | 7 | 4 | 2 | 5
Not completed — Death | 2 | 3 | 3 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 2
Not completed — Explant due to infection | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Medical reason | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Study site closure | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject non-compliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study completion | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Diabetic: This group contains all subjects that were enrolled and analyzed as part of the diabetic cohort.
- Idiopathic: This group contains all subjects that were enrolled and analyzed as part of the idiopathic cohort.
- Total: Total of all reporting groups
Arm/Group | Diabetic | Idiopathic | Total
Number analyzed (Participants) | 55 | 32 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 32 | 87
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.3 (9.8) | 39.4 (10.4) | 38.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 26 | 62
  Male | 19 | 6 | 25
Region of Enrollment [Number; unit: participants]
  United States | 55 | 32 | 87

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Frequency of Weekly Vomiting Episodes When the Device is Turned ON, Relative to When the Device is Turned OFF
Description: Diaries were used to record daily vomiting episodes for 28 days prior to each office follow-up visit. The weekly vomiting frequency (WVF) was based on the average number of weekly vomiting episodes recorded in the patient diary. The percent reduction is calculated as ((WVF during OFF - WVF during ON)/ (WVF during OFF))*100%. A positive reduction represents an improvement in WVF when the device was ON.
Time Frame: 4.5 months and 7.5 months
Population: The analysis population included subjects who were randomized, completed the study through the end of the blinded crossover period and provided evaluable measurements.
Measure: Median (Full Range); unit: percent reduction in WVF
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 32 | 20
percent reduction in WVF | 0 [-300 to 100] | 17.3 [-450 to 100]
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: There was no change in the frequency of weekly vomiting episodes from when stimulation was turned OFF to when stimulation was turned ON, µ = 0; Alternative hypothesis: There was a change in frequency of weekly vomiting episodes from when stimulation was turned OFF to when stimulation was turned ON, µ ≠ 0; Test type: Superiority or Other; p = 0.215, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons

2. Secondary Outcome: Percent Reduction in Symptom Score When the Device is Turned ON, Relative to When the Device is Turned OFF
Description: A symptom interview was conducted at each visit to assess vomiting, nausea, early satiety, bloating, postprandial fullness, epigastric pain and epigastric burning. The scale for each symptom ranges from 0 to 4, with 0 being absence of symptoms and 4 being extremely frequent (≥ 7 episodes per week). Total symptom score (TSS) is the sum of the individual frequency symptom scores. The percent reduction is calculated as ((TSS during OFF - TSS during ON)/ (TSS during OFF))*100%. A positive reduction represents an improvement in TSS when the device was ON.
Time Frame: 4.5 months and 7.5 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent reduction in symptom score
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 36 | 21
Percent reduction in symptom score | 0 [-250 to 100] | 0 [-87.5 to 100]
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: There was no change in total symptom score from when stimulation was turned OFF to when stimulation was turned ON, µ = 0; Alternative hypothesis: There was a change in total symptom score from when stimulation was turned OFF to when stimulation was turned ON, µ ≠ 0; Test type: Superiority or Other; p = 0.903, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.932, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons

3. Secondary Outcome: Percent Reduction in the Frequency of Weekly Vomiting Episodes at 12 Months Compared to Baseline
Description: Diaries were used to record daily vomiting episodes for 28 days prior to each office follow-up visit. The weekly vomiting frequency (WVF) was based on the average number of weekly vomiting episodes recorded in the patient diary. The percent reduction is calculated as ((WVF at baseline - WVF at 12 months)/ (WVF at baseline))*100%. A positive reduction represents an improvement in WVF at 12 months.
Time Frame: baseline and 12 months
Population: The analysis population included subjects who were randomized, completed the study at 12 months and provided evaluable measurements.
Measure: Median (Full Range); unit: Percent reduction in WVF
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 36 | 18
Percent reduction in WVF | 67.8 [-114.9 to 100] | 87.1 [-80.4 to 100]
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: There was no change from baseline in the long-term frequency of weekly vomiting episodes, µ = 0; Alternative hypothesis: There was a change from baseline in the long-term frequency of weekly vomiting episodes, µ ≠ 0; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons

4. Other Pre Specified Outcome: Percentage of Responders at 12 Months
Description: Responders were defined as having a 50% or greater reduction of WVF from baseline to 12 months. The percentage of responders was estimated as the proportion of the responders among all subjects who finished the 12-month visit. The percentage of responders was tested to determine if it was statistically greater than 50%.
Time Frame: baseline and 12 months
Population: as for outcome 3
Measure: Number; unit: Percentage of responders
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 36 | 18
Percentage of responders | 69 | 94
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: The percentage of responders was less than or equal to 50%; Alternative hypothesis: The percentage of responders was greater than 50%; Test type: Superiority or Other; p = 0.014, binomial, 1 sided — A one-sided significance level of 0.025 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, binomial, 1 sided — A one-sided significance level of 0.025 was applied to the test. No adjustments were made for multiple comparisons

5. Other Pre Specified Outcome: Change in Symptom Score at 12 Months Compared to Baseline.
Description: A symptom interview was conducted at each visit to assess vomiting, nausea, early satiety, bloating, postprandial fullness, epigastric pain and epigastric burning. The scale for each symptom ranges from 0 to 4, with 0 being absence of symptoms and 4 being extremely frequent (≥ 7 episodes per week). Total symptom score (TSS) is the sum of the individual frequency symptom scores. The change is calculated as TSS at baseline - TSS at 12 months. A positive change represents an improvement in TSS at 12 months.
Time Frame: baseline and 12 months
Population: The analysis population included subjects who were randomized and completed the study at 12 months.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 39 | 19
Scores on a scale | 6.79 (8.05) | 8.74 (7.46)
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: There was no change in total symptom score from baseline to 12 months, µ = 0; Alternative hypothesis: There was a change in total symptom score from baseline to 12 months, µ ≠ 0; Test type: Superiority or Other; p < 0.001, Paired t-test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons

6. Other Pre Specified Outcome: Change in Quality of Life (QOL) at 12 Months Compared to Baseline (Physical Component Summary)
Description: The QOL scores were collected using the SF-36 questionnaire, which included the scores in the following domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health. The raw score of 0 represents poor health and 100 represents best health. The physical component summary (PCS) score is a norm based score calculated from the raw scores of these 8 domains with a focus on physical health. The change in PCS is calculated as PCS at baseline - PCS at 12 months. A negative change in PCS represents an improvement in QOL.
Time Frame: baseline and 12 months
Population: The analysis population included subjects who were randomized and completed the study at 12 months.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 32 | 20
Scores on a scale | -6.9 (8.97) | -5.2 (10.43)
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: There was no change in PCS score from baseline to 12 months, µ = 0; Alternative hypothesis: There was a change in PCS score from baseline to 12 months, µ ≠ 0; Test type: Superiority or Other; p < 0.001, Paired t-test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.043, Paired t-test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons

7. Other Pre Specified Outcome: Change in Quality of Life at 12 Months Compared to Baseline (Mental Component Summary)
Description: The QOL scores were collected using the SF-36 questionnaire, which included the scores in the following domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health. The raw score of 0 represents poor health and 100 represents best health. The mental component summary (MCS) score is a norm based score calculated from the raw scores of these 8 domains with a focus on mental health. The change in MCS is calculated as MCS at baseline - MCS at 12 months. A negative change in MCS represents an improvement in QOL.
Time Frame: baseline and 12 months
Population: The analysis population included subjects who were randomized and completed the study at 12 months.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 39 | 19
Scores on a scale | -6.81 (15.15) | -7.15 (7.75)
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: There was no change in MCS score from baseline to 12 months, µ = 0; Alternative hypothesis: There was a change in MCS score from baseline to 12 months, µ ≠ 0; Test type: Superiority or Other; p = 0.009, Paired t-test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.001, Paired t-test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons

8. Other Pre Specified Outcome: Change in Gastric Emptying Results at 12 Months Compared to Baseline (2 Hours)
Description: Gastric emptying was evaluated using a standardized scintigraphy method and a low fat egg substitute test meal. After standard meal and marker preparation, the subsequent images were taken at 2 hours and 4 hours and percentage of gastric retention was evaluated. Change in 2-hour GET is calculated as % of gastric retention at 2 hours at baseline - % of gastric retention at 2 hours at 12 months. A positive change represents an improvement in gastric emptying at 12 months.
Time Frame: baseline and 12 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Percent retention
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 28 | 16
Percent retention | 18 [11 to 37.5] | 17.5 [-0.5 to 31]
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: There was no change in 2-hour gastric emptying from baseline to 12 months, µ = 0; Alternative hypothesis: There was a change in 2-hour gastric emptying from baseline to 12 months, µ ≠ 0; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons

9. Other Pre Specified Outcome: Change in Gastric Emptying Results at 12 Months Compared to Baseline (4 Hours)
Description: Gastric emptying was evaluated using a standardized scintigraphy method and a low fat egg substitute test meal. After standard meal and marker preparation, the subsequent images were taken at 2 hours and 4 hours and percentage of gastric retention was evaluated. Change in 4-hour GET is calculated as % of gastric retention at 4 hours at baseline - % of gastric retention at 4 hours at 12 months. A positive change represents an improvement in gastric emptying at 12 months.
Time Frame: baseline and 12 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Percent retention
Arm/Group | Diabetic | Idiopathic
Number analyzed (Participants) | 28 | 16
Percent retention | 22 [7.5 to 39.5] | 13.5 [-11 to 17]
Statistical Analysis 1: Comparison: Diabetic; Null hypothesis: There was no change in 4-hour gastric emptying from baseline to 12 months, µ = 0; Alternative hypothesis: There was a change in 4-hour gastric emptying from baseline to 12 months, µ ≠ 0; Test type: Superiority or Other; p = 0.016, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Idiopathic; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.236, Wilcoxon Signed Rank Test — A significance level of 0.05 was applied to the test. No adjustments were made for multiple comparisons

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study beginning at the time of patient enrollment until discontinuation from the study.
Description: All adverse events collected in the study were categorized by the investigator and reviewed by an adverse events commitee for causality. Tables below include all events that were classified as device-related, therapy-related, or undetermined. Events determined to be related to the patient's underlying condition (patient-related) are not included.
Arm/Group | Diabetic | Idiopathic
Serious Adverse Events (participants affected / at risk) | 8/55 | 4/32
Other Adverse Events (participants affected / at risk) | 13/55 | 9/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetic (N=55) | Idiopathic (N=32)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
High lead impedance (General disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Lead migration/dislodgment (General disorders) | 1 (2) | 1 (1)
Migration of implant (General disorders) | 1 (2) | 0 (0)
Neurostimulator migration (General disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetic (N=55) | Idiopathic (N=32)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Lead impedance NOS or high lead impedance (General disorders) | 11 (11) | 6 (7)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Early termination of the study impacted the ability to analyze the primary endpoint and secondary endpoint 1 for the idiopathic arm of the study. The minimum sample size for analysis of these endpoints was 32 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less